CLINICAL TRIAL: NCT01943318
Title: Prospective Cohort Study to Evaluate Long-term Outcomes in Patients With Liver Cirrhosis of Boramae Hospital
Brief Title: Boramae Hospital Liver Cirrhosis Patient Cohort Study
Status: Completed | Type: Observational
Sponsor: Seoul National University Boramae Hospital (Other)
Responsible Party: Principal Investigator, Won Kim, MD, PhD, Seoul National University Boramae Hospital
Other Study IDs: BRM_LC_Cohort
Record Dates: First submitted 2013-08-22; First posted 2013-09-16 (Estimated); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Liver Cirrhosis; Hepatocellular Carcinoma
Keywords: Liver Cirrhosis; Hepatocellular carcinoma
MeSH Terms: conditions — Liver Cirrhosis; Carcinoma, Hepatocellular | interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples With DNA — At enrollement, 20 ml of blood will be collected for freezing and storage of serum and plasma, and constitution of a DNA library
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (7):
- Alcohol: Alcoholic Liver Cirrhosis
  Participants will undergo liver biopsy. Participants will undergo hepatic venous pressure gradient measurement.
  Interventions: Procedure: Liver biopsy; Device: Hepatic venous pressure gradient (HVPG) measurement
- Hepatitis B virus: Hepatitis B virus (HBV) Liver Cirrhosis
  Interventions: Procedure: Liver biopsy; Device: Hepatic venous pressure gradient (HVPG) measurement
- Hepatitis C virus: Hepatitis C virus (HCV) Liver Cirrhosis
  Interventions: Procedure: Liver biopsy; Device: Hepatic venous pressure gradient (HVPG) measurement
- Autoimmune: Autoimmune Cirrhosis
  Interventions: Procedure: Liver biopsy; Device: Hepatic venous pressure gradient (HVPG) measurement
- Biliary: Primary or secondary biliary cirrhosis
  Interventions: Procedure: Liver biopsy; Device: Hepatic venous pressure gradient (HVPG) measurement
- Toxic: Medication related cirrhosis
  Interventions: Procedure: Liver biopsy; Device: Hepatic venous pressure gradient (HVPG) measurement
- Others: Hepatic venous pressure gradient (HVPG) measurement
  Interventions: Procedure: Liver biopsy; Device: Hepatic venous pressure gradient (HVPG) measurement

INTERVENTIONS:
Procedure: Liver biopsy — Histologic evaluation
Device: Hepatic venous pressure gradient (HVPG) measurement — Hepatic venous pressure gradient (HVPG) measurement

SUMMARY:
Liver cirrhosis represents a worldwide health problem and is a major cause of mortality. Cirrhosis is the common end for chronic alcohol abuse and hepatitis C and B virus infections. Patients who have cirrhosis have varying degrees of compensated liver function, and clinicians need to differentiate between those who have stable, compensated cirrhosis and those who have decompensated cirrhosis. It is shown various complications: portal hypertension, hepatocellular carcinoma, hepato-renal syndrome, etc.

Thus, it is important to have this information to manage disease and determine specific therapy. However, register-based studies in have not been reported in Korea.

The goal of this study is to describe the natural history of a large number of patients with liver cirrhosis prospectively followed, and to identify predictors of the occurrence of Hepatocellular carcinoma.

DETAILED DESCRIPTION:
The investigators are planning to recruit patients with liver cirrhosis, and collect the baseline clinical laboratory data. Biological tests, endoscopy,liver ultrasonography (including ARFI) and hepatic venous pressure gradient measurements will be performed if not done within 90 days prior to inclusion. During this visit, 20 ml of blood will be collected for freezing and storage of serum and plasma, and constitution of a DNA library.

Monitoring: Patients will have regular surveillance with blood test, liver ultrasonography and medical consultation at least every 6 months, periodic assessment of esophageal, gastric varices and portal hypertensive gastropathy (every 1 year) and prevention of their rupture if any. An additional blood sampling of 20 ml will be taken at baseline and every year in order to perform whole blood, serum, plasma, peripheral blood mononuclear cells and DNA libraries; Data will be standardized and centralized in a single database.

And alcoholic liver cirrhosis patients will undergo liver biopsy for polymerase chain reaction, western blot, immunohistochemistry and RNA analysis.

After measurement of hepatic venous pressure gradient and liver stiffness at baseline a non-selective beta-blocker (NSBB,carvedilol) was initiated and increased stepwise (weekly) until the systolic blood pressure remained at>100 mmHg and the heart rate was not <60. The maximum target dose for carvedilol 25 mg/day. The hepatic venous pressure gradient response to NSBB was again assessed 6 weeks after the intake of carvedilol. A hemodynamic response to NSBB treatment was defined as a reduction in hepatic venous pressure gradient >=20% compared to baseline or to an absolute value <=12 mmHg. Compliance with therapy was monitored by monitoring of heart rate and blood pressure during clinical visits.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥19years old Proven cirrhosis
* No previous hepatocellular carcinoma (treated or not)
* Signed informed consent

Exclusion Criteria:

* serious associated short-term life threatening disease (except associated HIV viral infection and the liver disease itself)
* liver focal lesion suggestive of hepatocellular carcinoma
* patient under guardianship
* pregnant women
* inability to regular monitoring, for whatever reason

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Seoul National University Boramae hospital
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2022-05 (Actual); Study Completion 2022-05 (Actual)

PRIMARY OUTCOMES:
Liver-related outcome: Decompensated liver cirrhosis (ascites, variceal bleeding, hepatic encepahlopathy), occurence of hepatocellular carcinoma | 5 years
  Cumulative incidence within 5 years Laboratory Tests: Albumin, Total bilirubin, prothrombin time, Platelet Hepatic venous pressure gradient measurement Imaging study like Liver CT or Liver ultrasonography Endoscopy for varix evaluation

SECONDARY OUTCOMES:
Mortality | 5 years
  overall mortality - whatever the cause of death
Liver-related mortality | 5 years
  cumulative incidence of liver-related deaths

CONTACTS AND LOCATIONS:
Overall Officials: Won Kim, MD, Principal Investigator — Boramae Hospital
Locations (1):
- SNU-SMG Boramae Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dam Fialla A, Schaffalitzky de Muckadell OB, Touborg Lassen A. Incidence, etiology and mortality of cirrhosis: a population-based cohort study. Scand J Gastroenterol. 2012 Jun;47(6):702-9. doi: 10.3109/00365521.2012.661759. Epub 2012 Mar 19. PMID 22428859
- [Background] Reiberger T, Ferlitsch A, Payer BA, Pinter M, Homoncik M, Peck-Radosavljevic M; Vienna Hepatic Hemodynamic Lab. Non-selective beta-blockers improve the correlation of liver stiffness and portal pressure in advanced cirrhosis. J Gastroenterol. 2012 May;47(5):561-8. doi: 10.1007/s00535-011-0517-4. Epub 2011 Dec 15. PMID 22170417
- [Derived] Cho Y, Choi YI, Oh S, Han J, Joo SK, Lee DH, Jung YJ, Kim BG, Lee KL, Kim W. Point shear wave elastography predicts fibrosis severity and steatohepatitis in alcohol-related liver disease. Hepatol Int. 2020 Mar;14(2):270-280. doi: 10.1007/s12072-019-10009-w. Epub 2019 Dec 19. PMID 31858403
- [Derived] Kim HY, So YH, Kim W, Ahn DW, Jung YJ, Woo H, Kim D, Kim MY, Baik SK. Non-invasive response prediction in prophylactic carvedilol therapy for cirrhotic patients with esophageal varices. J Hepatol. 2019 Mar;70(3):412-422. doi: 10.1016/j.jhep.2018.10.018. Epub 2018 Oct 31. PMID 30389550